CLINICAL TRIAL: NCT06285981
Title: Observational Retrospective Study to Assess the Clinical Benefit and Safety Profile of the Intramedullary Nail CHIMAERA in Adult Patient Who Have Suffered Pertrochanteric, Intertrochanteric and Subtrochanteric Fractures of the Femur in Daily Practice: CHIMAERA Study
Brief Title: Retrospective Study Chimaera Long Nail in Adult Patient
Status: Completed | Type: Observational
Sponsor: Orthofix s.r.l. (Industry)
Responsible Party: Sponsor
Other Study IDs: OCI_2206
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Results first posted 2025-08-07 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Pertrochanteric Fracture of Femur; Intertrochanteric Fracture of Femur; Subtrochanteric Fracture of Femur
Keywords: intramedullary nail; chimaera; orthofix; fractures; femur
MeSH Terms: conditions — Hip Fractures; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients with femur fractures: adult patients with pertrochanteric, intertrochanteric and subtrochanteric fractures of the femur
  Interventions: Device: Chimaera Long Nail

INTERVENTIONS:
Device: Chimaera Long Nail — The CHIMAERATM, is an internal fixation system intended intended for insertion into the medullary canal of a femur in individuals suffering from stable and unstable pertrochanteric, intertrochanteric and subtrochanteric fractures of the femur alone or when these fractures occur in combination with shaft fractures extending distally to a point approximately 10cm proximal to the intercondylar notch.

SUMMARY:
The CHIMERA study intends to evaluate the clinical benefits of the study medical device in the standard clinical practice.

DETAILED DESCRIPTION:
The CHIMERA study intends to evaluate the clinical benefits of the study medical/investigational device in the standard clinical practice. The study will be conducted in two sites located in Italy; both considered reference sites for the treatment of adult patients with pertrochanteric, intertrochanteric and subtrochanteric fractures of the femur, where the usage of Orthofix® Chimaera Hip Fracture SystemTM (from now on CHIMAERA) was part of the normal clinical practice. The CHIMAERA, is an internal fixation system intended for insertion into the medullary canal of a femur in individuals suffering from stable and unstable pertrochanteric, intertrochanteric and subtrochanteric fractures of the femur alone or when these fractures occur in combination with shaft fractures extending distally to a point approximately 10cm proximal to the intercondylar notch. The participant investigators will retrospectively include a maximum of 44 patients meeting inclusion and exclusion criteria (considering an imprecision of 5%) that will contribute for approximately 44 patients in which CHIMAERA was used.

The study is designed to analyze medical records of adult patients who underwent CHIMAERA implantation from 2018 to 2023 in the standard clinical practice setting.

ELIGIBILITY:
Inclusion Criteria:

1. The patient expressed his willingness to participate in the Study by signing and dating informed consent.
2. Patients who had a regular indication for surgical intervention with the long variant of CHIMAERATM according to the manufacturer's IFU.
3. Patients equal or older than 18 years at the time of surgery.
4. Patients who underwent surgery performed with CHIMAERATM.
5. Patients with clinical data registered in her/his medical records sufficient to assess the safety and efficacy endpoints of the study.

Exclusion Criteria:

1. Patient who had/has a medical condition that is a contraindication according to the manufacturer's IFU leaflet.
2. Patient has been diagnosed with bilateral proximal femur fractures.
3. Patient who needed the application of, or ha already in-situ a concomitant not permitted device which cannot be safely removed.
4. Patient with other concurrent medical or non-medical condition that in the opinion of the participating investigator may prevent participation or otherwise render the patient ineligible for the study.
5. The patient is participating in other clinical studies, or he/she has participated in other clinical studies in the 3 months prior signing the informed consent .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults suffering from pertrochanteric, intertrochanteric and subtrochanteric fractures of the femur, where the usage of Orthofix® Chimaera Hip Fracture SystemTM (from now on CHIMAERATM) was part of the normal clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - AORN Sant'Anna e San Sebastiano, Caserta, CE
  - Craeggi Hospital, Florence, FI

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients With Femur Fractures
Started | 44
Completed | 44
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Femur Fractures
Number analyzed (Participants) | 44
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 74 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 44
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients in Which Bone Union Has Been Achieved
Description: The clinical benefit of CHIMAERATM will be assessed by the percentage of patients in which bone union has been achieved within 12 months from the nail implant.
Time Frame: 12 months
Population: Only 42 out of 44 enrolled patient were analysed for the performance endpoint because Two patients did not meet the CIP criteria for the primary endpoint evaluation and were not included in the efficacy analysis of clinical benefit, but were included in study evaluation for safety.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Femur Fractures
Number analyzed (Participants) | 42
Participants | 42

2. Secondary Outcome: Percent of Patients That Required a Reoperation
Description: The safety profile of CHIMAERATM will be assessed through the percentage of patients that required a reoperation (i.e., additional surgery).
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Femur Fractures
Number analyzed (Participants) | 44
Participants | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Patients With Femur Fractures
All-Cause Mortality (participants affected / at risk) | 0/44
Serious Adverse Events (participants affected / at risk) | 2/44
Other Adverse Events (participants affected / at risk) | 2/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Femur Fractures (N=44)
Deep infection (Infections and infestations) | 1 (1) — Deep infection not dependent on nail, but on patient's physical condition. nail removal plus antibiotic therapy still ongoing at end of infection, will need to undergo another procedure.
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — Patient underwent reduction and synthesis procedure for femoral shaft fracture with plate and screws plus bank bone stick with cerclage
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Femur Fractures (N=44)
Covid Infection (Infections and infestations) | 1 (1)
Anemia (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-07-13): https://cdn.clinicaltrials.gov/large-docs/81/NCT06285981/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-06): https://cdn.clinicaltrials.gov/large-docs/81/NCT06285981/SAP_001.pdf